CLINICAL TRIAL: NCT00876876
Title: International, Multicenter, Open-Label and Randomized Withdrawal Study of Oral Lixivaptan in Heart Failure Patients With Chronic Hyponatremia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Created Extension study - This study was no longer feasible
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cesare Orlandi, MD, Cardiokine Biopharma, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CK-LX3422
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Hypervolemic Hyponatremia
Keywords: hypervolemic hyponatremia; serum sodium; fluid overload; heartfailure; acute heart failure; vasopressin antagonist
MeSH Terms: conditions — Edema | interventions — lixivaptan

ARMS (2):
- Placebo QD or BID (Placebo Comparator): Placebo QD or BID
  Interventions: Drug: Lixivaptan
- Lixivaptan QD or BID (Experimental): Lixivaptan QD or BID
  Interventions: Drug: Lixivaptan

INTERVENTIONS:
Drug: Lixivaptan — Capsules containing 25, or 50 mg doses of oral lixivaptan to be administered BID or QD Lixivaptan will be administered for 12 weeks in the Open-Label Period which will be followed by a 4 week Randomized, Placebo-Controlled period.

SUMMARY:
To demonstrate that after 12 weeks of open-label lixivaptan treatment, serum sodium is maintained in hyponatremic patients continuing to receive lixivaptan compared to placebo during the 4 week double blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women with age greater than or equal to 18 years.
2. Prior successful participation in a randomized, blinded, placebo-controlled Phase 3 lixivaptan study of hyponatremia in Heart Failure (Protocol CK-LX3401) with evidence of continued need for therapy as follows:

   * Patient completed full course of treatment (e.g., either placebo or lixivaptan). Treatment assignments for Protocol CK-LX3401 will not be unblinded prior to participation in the extension study.
   * Baseline serum sodium concentration < 135 mEq/L following a 30 day post treatment follow-up period in a lixivaptan hyponatremia parent trial. Repeat measures of serum sodium are allowed; the last serum sodium result within 24 hours prior to randomization will serve as the qualifying measurement.
3. The patient has clinical evidence of volume overload with at least one of the following:

   * Dyspnea
   * Pulmonary congestion (rales)
   * Peripheral edema
   * Increased jugular venous pressure and/or hepatic congestion with ascites
   * Chest x-ray consistent with CHF; OR
   * Plasma BNP ≥150 pg/mL or NT pro-BNP ≥ 450 pg/mL

Exclusion Criteria:

1. Women who are pregnant (positive pregnancy test), breastfeeding or who will not adhere to the reproductive precautions as outlined in this protocol and in the informed consent form.
2. Inability to provide informed consent.
3. Acute severe hyponatremia with overt symptoms of hyponatremia requiring immediate medical intervention (e.g., coma, seizures).
4. Acute or transient hyponatremia (e.g., associated with head trauma or postoperative state).
5. Hyponatremia in hypovolemic states. Hypovolemia is defined as the presence of clinical evidence of fluid volume depletion.
6. Euvolemic Hyponatremia (e.g., SIADH, etc.). Euvolemic hyponatremia is defined as low serum sodium in the presence of normal total body sodium due to mild to moderate increases in total body water without edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that after 12 weeks of open-label lixivaptan treatment, serum sodium is maintained in hyponatremic patients continuing to receive lixivaptan compared to placebo during the 4 week double blind treatment period. | 12 weeks

SECONDARY OUTCOMES:
To demonstrate that after 12 weeks of open-label lixivaptan treatment, improvements in the time to complete the Trail Making Test (Part B) will be maintained in patients continuing to receive lixivaptan. | 20 weeks